CLINICAL TRIAL: NCT04492137
Title: Prospective Comparison Between Ultra Early NKF Versus Standard Cannulation Alone in a Group of High and Low Risk of Pep, Submitted to Pep Prophylaxis
Brief Title: Prospective Comparison Between Ultra Early NKF Versus Standard Cannulation Alone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Minho (Other)
Collaborators: Unidade Local de Saúde do Alto Minho (Other)
Responsible Party: Principal Investigator, Luis Lopes, Assistant Professor (MD, PhD, MBA), University of Minho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 32/2020
Record Dates: First submitted 2020-07-09; First posted 2020-07-30 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Pancreatitis
Keywords: ERCP; Biliary cannulation; Needle-knife fistulotomy; Standard cannulation methods
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: We will conduct a prospective randomized study. Participants will be randomized by computer into two groups at a 1:1 ratio
  1. participants submitted to ultra early NKF
  2. participants submitted to standard cannulation techniques (including double-guidewire-assisted cannulation)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra Early NKF group (Experimental): Patients submitted to Ultra early NKF in a consecutive fashion by an expert endoscopist
  Interventions: Procedure: Cannulation technique
- Standard cannulation techniques group (including double-guidewire-assisted cannulation) (No Intervention): Patients submitted to standard cannulation techniques (including double-guidewire-assisted cannulation) in a consecutive fashion by an expert endoscopist

INTERVENTIONS:
Procedure: Cannulation technique — Participants in the ultra early NKF group will be submitted to 2 standard cannulation attempts (2 contacts with the papilla) before starting NKF. If any of these 2 attemps is successful, NKF won't take place. If NKF is indeed performed and cannulation is not achieved within 8 minutes, the endoscopist is free to perform techniques other than NKF. On the other hand, participants in the standard cannulation group in which cannulation is not achieved within 8 minutes can cross-over to other advanced cannulation techniques (e.g. NKF). For ethical reasons we choose to exclude flat and intradiverticular/diverticular border papillas.
  During ERCP all participants will be submitted to PEP prophylaxis with rectal indomethacin. A pancreatic stent will be placed whenever there is cannulation or opacification of the Wirsung duct.
  For the purposes of the study, a dedicated form (attached) will be created with the various variables to be analyzed
  Arms: Ultra Early NKF group

SUMMARY:
Compare the ultra early fistulotomy strategy with standard cannulation methods for accessing the bile duct during endoscopic retrograde cholangiopancreatography (ERCP)

DETAILED DESCRIPTION:
1. Introduction

   Endoscopic retrograde cholangiopancreatography (ERCP) is an advanced procedure which is widely used in the diagnosis and treatment of a variety of benign and malignant pancreatobiliary disorders1,2,3,4,5.

   Selective cannulation of the common bile duct (CBD) is the most important and challenging step in a biliary endoscopic retrograde cholangiopancreatography6,7. However, in the first ERCP, even in experienced hands, biliary cannulation may fail in up to 15 % - 35 % of cases when using standard methods alone8. In this subset of patients, additional cannulation techniques are needed to access the CBD in order to continue with the ERCP.

   Precut is the most common strategy used by experienced endoscopists, when conventional methods have failed7. Needle knife fistulotomy (NKF) and conventional precut are the two most common variants. Recently published guidelines recommend opting for NKF, as evidence suggests a lower risk of adverse events, especially pancreatitis, when used early in the biliary cannulation algorithm7,9.

   Technically NKF is the creation of an artificial fistula between the most protuberant portion of the papilla, which represents the intraduodenal portion of the CBD and the biliary tract by using a diathermic cutter of the needle type6,10,11,12,13,14,15,16,17,18. Its big advantage over conventional precut is that it avoids the contact of the cutting device with the papillary orifice and therefore avoiding direct thermal injury to the pancreatic duct.

   Although NKF was originally developed as a rescue technique, to be used after previous failed standard cannulations attempts, it is being increasingly used at an early stage during ERCP. Given its safety and feasibility some authors even advocate, the once unreasonable, primary use without previous standard cannulation attempts10,11,19,20.
2. Financial resources

   All participants included in this study will perform ERCP, laboratory tests and other complementary diagnostic tests after a duly justified medical prescription. Therefore there are no additional costs or consumption of hospital resources.
3. Ethical considerations In this study, participants will be included after informed consent. Anonymity and confidentiality will be safeguarded by assigning an individual numeric code. It will also be explained the possibility of withdrawing from the study at any time, with the guarantee of the total elimination of data. All researchers involved in the study will adhere to the Rules of Ethical Conduct and Best Practices in order to comply with the precepts of the Declaration of Helsinki, the Convention on Human Rights and Biomedicine, the guidelines of the Council for International Organizations of Medical Sciences and the Guide to Good Clinical Practice.
4. Statistical analysis

   Qualitative variables will be summarized using absolute and relative frequencies, and quantitative variables will be summarized using the mean and standard deviation or the median and interquartile range, depending on their distribution profiles. The normality of the quantitative variables will be assessed using the histogram distribution.

   A sample of 334 (167 in each group) patients will provide 80% power to detect a difference of 5% in pancreatitis rates between the two groups based on a chi-square test, assuming a pancreatitis rate of 1% among primary fistulotomy, 6 and a one-tailed alpha of 0.05.

   Relations between categorical variables will be assessed using a chi-square test and Fisher´s exact test. Differences between two or more groups of independent non-normally distributed quantitative variables will be evaluated using a Kruskal-Wallis test.

   To explain the risk of pancreatitis, a binomial logistic regression model with multiple predictors will be performed.

   The null hypothesis will be rejected when the test statistics p-values are less than <0.05. Statistical analysis, sample size calculation and graphics will be performed using Stata software (StataCorp. 2015. Stata Statistical Software: Release 14. College Station, StataCorp LP)
5. Expected results

The results of this study will contribute to a better understanding of what is the best algorithm to follow when performing an ERCP.

ELIGIBILITY:
From June 1, 2020 to June 1, 2022, all individuals referred for ERCP in the Digestive Endoscopy Unit of Santa Luzia Hospital (Unidade Local de Saúde do Alto Minho) will be invited to participate in the study.

Inclusion Criteria:

* ERCP with indication for biliary access
* Naïve papilla

Exclusion Criteria:

* Flat papillas
* Intradiverticular / Diverticular border papillas
* Patients unable to sign or understand the informed consent
* Patients with surgically altered anatomy
* Patients with tumors of the papilla
* Previous sphincterotomy
* Spontaneous papillary fistula
* Papilla not visualized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 30 days from the procedure
  Comparison of adverse event rate between the two strategies
Technical success | 1 day (same day of the procedure)
  Comparison of technical success between the two strategies

SECONDARY OUTCOMES:
Adverse event rate among sub groups | 30 days from the procedure
  Comparison of adverse event rate among sub groups (high and low risk of pancreatitis)
Technical success among sub groups | 1 day (same day of the procedure)
  Comparison of technical success rate among sub groups (high and low risk of pancreatitis)

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Luzia Hospital, ULS Alto Minho, Viana do Castelo, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canena J, Liberato M, Coutinho AP, Marques I, Romao C, Veiga PM, Neves BC. Predictive value of cholangioscopy after endoscopic management of early postcholecystectomy bile duct strictures with an increasing number of plastic stents: a prospective study (with videos). Gastrointest Endosc. 2014 Feb;79(2):279-88. doi: 10.1016/j.gie.2013.07.022. Epub 2013 Sep 5. PMID 24012251
- [Background] Canena J, Coimbra J, Carvalho D, Rodrigues C, Silva M, Costa M, Horta D, Mateus Dias A, Seves I, Ramos G, Ricardo L, Coutinho AP, Romao C, Veiga PM. Endoscopic bilio-duodenal bypass: outcomes of primary and revision efficacy of combined metallic stents in malignant duodenal and biliary obstructions. Dig Dis Sci. 2014 Nov;59(11):2779-89. doi: 10.1007/s10620-014-3199-y. Epub 2014 May 13. PMID 24821464
- [Background] Canena J, Liberato M, Meireles L, Marques I, Romao C, Coutinho AP, Neves BC, Veiga PM. A non-randomized study in consecutive patients with postcholecystectomy refractory biliary leaks who were managed endoscopically with the use of multiple plastic stents or fully covered self-expandable metal stents (with videos). Gastrointest Endosc. 2015 Jul;82(1):70-8. doi: 10.1016/j.gie.2014.11.038. Epub 2015 Mar 11. PMID 25771064
- [Background] Canena J. Once upon a Time a Guideline Was Used for the Evaluation of Suspected Choledocholithiasis: A Fairy Tale or a Nightmare? GE Port J Gastroenterol. 2018 Jan;25(1):6-9. doi: 10.1159/000481688. Epub 2017 Nov 8. No abstract available. PMID 29457044
- [Background] Canena J, Lopes L, Fernandes J, Alexandrino G, Lourenco L, Libanio D, Horta D, Giestas S, Reis J. Outcomes of Single-Operator Cholangioscopy-Guided Lithotripsy in Patients with Difficult Biliary and Pancreatic Stones. GE Port J Gastroenterol. 2019 Mar;26(2):105-113. doi: 10.1159/000488508. Epub 2018 May 16. PMID 30976615
- [Background] Lopes L, Dinis-Ribeiro M, Rolanda C. Safety and efficacy of precut needle-knife fistulotomy. Scand J Gastroenterol. 2014 Jun;49(6):759-65. doi: 10.3109/00365521.2014.898085. Epub 2014 Mar 18. PMID 24641260
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Testoni PA, Testoni S, Giussani A. Difficult biliary cannulation during ERCP: how to facilitate biliary access and minimize the risk of post-ERCP pancreatitis. Dig Liver Dis. 2011 Aug;43(8):596-603. doi: 10.1016/j.dld.2011.01.019. Epub 2011 Mar 4. PMID 21377432
- [Background] Lopes L, Dinis-Ribeiro M, Rolanda C. Early precut fistulotomy for biliary access: time to change the paradigm of "the later, the better"? Gastrointest Endosc. 2014 Oct;80(4):634-641. doi: 10.1016/j.gie.2014.03.014. Epub 2014 May 6. PMID 24814775
- [Background] Jin YJ, Jeong S, Lee DH. Utility of needle-knife fistulotomy as an initial method of biliary cannulation to prevent post-ERCP pancreatitis in a highly selected at-risk group: a single-arm prospective feasibility study. Gastrointest Endosc. 2016 Nov;84(5):808-813. doi: 10.1016/j.gie.2016.04.011. Epub 2016 Apr 19. PMID 27102829
- [Background] Jang SI, Kim DU, Cho JH, Jeong S, Park JS, Lee DH, Kwon CI, Koh DH, Park SW, Lee TH, Lee HS. Primary Needle-Knife Fistulotomy Versus Conventional Cannulation Method in a High-Risk Cohort of Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis. Am J Gastroenterol. 2020 Apr;115(4):616-624. doi: 10.14309/ajg.0000000000000480. PMID 31913191
- [Background] Mavrogiannis C, Liatsos C, Romanos A, Petoumenos C, Nakos A, Karvountzis G. Needle-knife fistulotomy versus needle-knife precut papillotomy for the treatment of common bile duct stones. Gastrointest Endosc. 1999 Sep;50(3):334-9. doi: 10.1053/ge.1999.v50.98593. PMID 10462652
- [Background] Katsinelos P, Gkagkalis S, Chatzimavroudis G, Beltsis A, Terzoudis S, Zavos C, Gatopoulou A, Lazaraki G, Vasiliadis T, Kountouras J. Comparison of three types of precut technique to achieve common bile duct cannulation: a retrospective analysis of 274 cases. Dig Dis Sci. 2012 Dec;57(12):3286-92. doi: 10.1007/s10620-012-2271-8. Epub 2012 Jun 20. PMID 22714730
- [Background] Abu-Hamda EM, Baron TH, Simmons DT, Petersen BT. A retrospective comparison of outcomes using three different precut needle knife techniques for biliary cannulation. J Clin Gastroenterol. 2005 Sep;39(8):717-21. doi: 10.1097/01.mcg.0000173928.82986.56. PMID 16082283
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N. Effect of precut sphincterotomy on biliary cannulation based on the characteristics of the major duodenal papilla. Clin Gastroenterol Hepatol. 2007 Sep;5(9):1113-8. doi: 10.1016/j.cgh.2007.05.014. Epub 2007 Aug 6. PMID 17689295
- [Background] Lee TH, Bang BW, Park SH, Jeong S, Lee DH, Kim SJ. Precut fistulotomy for difficult biliary cannulation: is it a risky preference in relation to the experience of an endoscopist? Dig Dis Sci. 2011 Jun;56(6):1896-903. doi: 10.1007/s10620-010-1483-z. Epub 2010 Nov 17. PMID 21082346
- [Background] Harewood GC, Baron TH. An assessment of the learning curve for precut biliary sphincterotomy. Am J Gastroenterol. 2002 Jul;97(7):1708-12. doi: 10.1111/j.1572-0241.2002.05829.x. PMID 12135022
- [Background] Donnellan F, Zeb F, Courtney G, Aftab AR. Suprapapillary needleknife fistulotomy: a safe and effective method for accessing the biliary system. Surg Endosc. 2010 Aug;24(8):1937-40. doi: 10.1007/s00464-010-0881-9. Epub 2010 Feb 5. PMID 20135176
- [Background] Chen DD, Keswani RN. Is Needle Knife Fistulotomy a Shortcut to Preventing Postendoscopic Retrograde Pancreatitis? Am J Gastroenterol. 2020 Apr;115(4):535-536. doi: 10.14309/ajg.0000000000000553. PMID 32049681
- [Background] Khatibian M, Sotoudehmanesh R, Ali-Asgari A, Movahedi Z, Kolahdoozan S. Needle-knife fistulotomy versus standard method for cannulation of common bile duct: a randomized controlled trial. Arch Iran Med. 2008 Jan;11(1):16-20. PMID 18154417